CLINICAL TRIAL: NCT06755892
Title: The Effect of 16-week Dietary Intake of Food Supplements Containing Collagen on Dermis Density and Other Skin Parameters: Double Blind, Placebo-controlled, Randomised Five-way Study Comparing the Efficacy of Four Test Products
Brief Title: The Effect of 16-week Dietary Intake of Food Supplements Containing Collagen and MSM on Skin
Acronym: TO-COSKIN3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VIST - Faculty of Applied Sciences (Other)
Collaborators: Tosla d.o.o. (Industry); Slovenian Research and Innovation Agency (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VIST TO-COSKIN3 03-2024
Record Dates: First submitted 2024-12-24; First posted 2025-01-01 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-10

CONDITIONS: Dermis Density; Wrinkles; Dermis Thickness; Skin Texture; Skin Elasticity; Skin Redness
MeSH Terms: conditions — Erythema

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- IP1 group (Active Comparator): Participants will receive investigational product 1 containing collagen (5 g/ 25 mL), MSM (1.0 g/ 25 mL) and vitamin C (80 mg/ 25 mL) for 16 weeks.
  Interventions: Dietary Supplement: ColMSM-HL
- IP2 group (Active Comparator): Participants will receive investigational product 2 containing collagen (3 g/ 25 mL), MSM (1.5 g/ 25 mL) and vitamin C (80 mg/ 25 mL), 25 mL/daily for 16 weeks.
  Interventions: Dietary Supplement: ColMSM-LH
- IP3 group (Active Comparator): Participants will receive investigational product 3 containing collagen (3 g/ 25 mL), MSM (1.0 g/ 25 mL) and vitamin C (80 mg/ 25 mL), 25 mL/daily for 16 weeks.
  Interventions: Dietary Supplement: ColMSM-LL
- IP4 group (Active Comparator): Participants will receive investigational product 4 containing containing collagen (3 g/ 25 mL) and vitamin C (80 mg/ 25 mL), 25 mL/daily for 16 weeks.
  Interventions: Dietary Supplement: Col-L
- Placebo group (Placebo Comparator): Placebo group participants will receive placebo syrup without active ingredients (0 mg of collagen, 0 mg of MSM and 0 mg of vitamin C), 25 mL/daily for 16 weeks.
  Interventions: Dietary Supplement: Placebo syrup

INTERVENTIONS:
Dietary Supplement: ColMSM-HL — Participants will test continuous administration of investigational product for 16 weeks.
  Other Names: Investigational product 1
  Arms: IP1 group
Dietary Supplement: Placebo syrup — Participants will test continuous administration of placebo product for 16 weeks.
  Arms: Placebo group
Dietary Supplement: ColMSM-LH — Participants will test continuous administration of investigational product for 16 weeks.
  Other Names: Investigational product 2
  Arms: IP2 group
Dietary Supplement: ColMSM-LL — Participants will test continuous administration of investigational product for 16 weeks.
  Other Names: Investigational product 3
  Arms: IP3 group
Dietary Supplement: Col-L — Participants will test continuous administration of investigational product for 16 weeks.
  Other Names: Investigational product 4
  Arms: IP4 group

SUMMARY:
The aim of the study is to compare the effects of multiple-dose 16 weeks daily dietary supplementation with 5 g or 3 g of collagen in combination with 1 g or 1.5 g of MSM and 80 mg vitamin C (see 1.2. Investigational and placebo product profile) on skin in healthy human subjects in comparison to placebo product. The main objective is to show that test products have beneficial effects on dermis density, and also on other skin parameters and to investigate differences in the effects among test products.

DETAILED DESCRIPTION:
Single centre, randomized, double-blind, placebo-controlled, one-period effectiveness study will include 135 subjects. Subjects will be divided in five groups, 27 in each. Test group 1 (IP1 group) will receive investigational product 1 (IP1, daily dose 25 mL: collagen 5 g, MSM: 1,0 g, vitamin C: 80 mg), test group 2 (IP2 group) will receive investigational product 2 (IP2, daily dose 25 mL: collagen 3 g, MSM: 1,5 g, vitamin C: 80 mg), test group 3 (IP3 group) will receive investigational product 3 (IP3, daily dose 25 mL: collagen 3 g, MSM: 1,0 g, vitamin C: 80 mg), test group 4 (IP4 group will receive investigational product 4 (IP4, daily dose 25 mL: collagen 3 g, vitamin C: 80 mg) and the placebo group will receive placebo product without those active ingredients (25 mL: 0 g collagen, 0 g MSM). Participants will test continuous administration of placebo or investigational products for 16 weeks to demonstrate and assess multiple-dose effects.

ELIGIBILITY:
Inclusion criteria:

* Caucasian female volunteers aged between 40 and 65 years at the time of the signature of Informed consent form (ICF),
* Signed Informed consent form (ICF),
* Fitzpatrick skin phototypes I-IV,
* Signs of skin aging,
* In good general health condition,
* BMI < 35
* Willingness to avoid a consumption of any food supplements containing methylsulfonylmethane (MSM), antioxidants, collagen and other protein-based food supplements during the study,
* Willingness to follow all study procedures and keeping a diary during the study (to follow their compliance and palatability).
* Willingness to maintain their living habits and to not begin or change any oestrogen or progesterone therapies,
* Willingness to avoid shaving/depilation of their arms during the study,
* Willingness not to change cosmetic treatment routine during the study,
* Willingness to avoid rejuvenation treatments during the study.

Exclusion criteria:

* Pregnancy or breastfeeding,
* Known or suspected allergy to any ingredient of the tested products,
* Changes in dietary habits and dietary supplementation in the last three months prior to inclusion,
* Regular use of food supplements containing MSM, antioxidants, collagen or other protein-based food supplements in the last three months prior to inclusion,
* Veganism,
* Changes in cosmetic facial and body care routine in the last month prior to inclusion,
* Diagnosed and uncontrolled/untreated/unregulated disease,
* Any clinically significant history of serious metabolic disease, digestive tract disease, liver disease, kidney disease, haematological disease,
* Intake of drugs with any impact on skin reactions (e.g., glucocorticoids, antihistamines, and immunomodulators),
* Any clinically significant acute or chronic skin diseases,
* Skin pigmentation disorders on measuring sites,
* Anticipated sunbathing or solarium visits before or during the study,
* Invasive rejuvenation treatments (e.g. needle rollers, needle mesotherapy, deep/medium-deep chemical peels, laser therapy etc.) in the last 4 months prior to study entry,
* Non-invasive rejuvenation treatments (e.g. radiofrequency, electrotherapy, ultrasound, IPL therapy) in the last month prior to study entry,
* Shaving/depilation of the arms in the last 14 days before inclusion,
* Mental incapacity that precludes adequate understanding or cooperation.

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 139 (Actual)
Dates: Start 2025-01-27 (Actual); Primary Completion 2025-06-17 (Actual); Study Completion 2025-06-17 (Actual)

PRIMARY OUTCOMES:
Change of dermis density from baseline in all test groups in comparison to placebo group after 16 weeks of dietary supplementation | 16 weeks
  Significant change of dermis density from baseline in test groups, in comparison to placebo group after 16 weeks of dietary supplementation with study product is expected. Dermis density will be assessed through ultrasonographic dermis intensity measurement. Differences in change of dermis density between test groups under primary objective conditions will also be evaluated.

SECONDARY OUTCOMES:
Change of wrinkle volume from baseline in test groups, in comparison to placebo group after 16 weeks of dietary supplementation | 16 weeks
  Assessment of the effects of investigational product on periorbital wrinkles after 16 weeks of dietary supplementation will be done using topography measurements. Differences between test groups will also be evaluated.
Change of skin texture from baseline in test groups, in comparison to placebo group after 16 weeks of dietary supplementation | 16 weeks
  For assessments of skin texture topography roughness measurements (Ra) will be performed. Significant changes from baseline in test groups, in comparison to placebo group after 16 weeks of dietary supplementation is expected. Differences between test groups will also be evaluated.
Change of skin redness from baseline in test groups, in comparison to placebo group after 16 weeks of dietary supplementation | 16 weeks
  Assessment of the effects of the investigational product on skin redness after 16 weeks of dietary supplementation. Skin redness (redness score, variation and uniformity) will be measured using Antera 3D CS. Differences between test groups will also be evaluated.
Change of dermis thickness from baseline in test groups, in comparison to placebo group after 16 weeks of dietary supplementation | 12 weeks
  Significant change of dermis thickness from baseline in test group, in comparison to placebo group after 16 weeks of dietary supplementation with study product is expected. Dermis density will be assessed using ultrasonography. Differences between test groups will also be evaluated.
Change of skin elasticity from baseline in test groups, in comparison to placebo group after 16 weeks of dietary supplementation | 16 weeks
  Elasticity measurements will be performed. Significant changes from baseline in test groups in comparison to the placebo group after 16 weeks of dietary supplementation are expected. Differences between test groups will also be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Katja Žmitek, PhD, Study Director — Head of Reasearch Group
Locations (1):
- VIST - Faculty of Applied Sciences, Institute of Cosmetics, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No